CLINICAL TRIAL: NCT06899594
Title: A Pilot Study in North Louisiana to Assess the Tolerability of Psilocybin as Well as Its Capacity to Promote Abstinence From Methamphetamine
Brief Title: Psilocybin for Methamphetamine Addiction
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kevin Murnane (Other)
Responsible Party: Sponsor-Investigator, Kevin Murnane, Associate Professor, Louisiana State University Health Sciences Center Shreveport
Organization: Louisiana State University Health Sciences Center Shreveport (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002094
Record Dates: First submitted 2024-11-27; First posted 2025-03-28 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-03

CONDITIONS: Methamphetamine Use Disorder
Keywords: Methamphetamine; Psilocybin; Psychedelics; Methamphetamine Use Disorder; Stimulant Use Disorder; Methamphetamine Addiction; Addiction; Substance Use Disorder; Abstinence
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin (Experimental): Participants will be administered 25mg of Psilocybin.
  Interventions: Drug: Psilocybin 25 mg

INTERVENTIONS:
Drug: Psilocybin 25 mg — 25 mg administered orally (capsules)

SUMMARY:
The primary purpose of this study is to preliminarily determine if the use of psilocybin to promote abstinence from methamphetamine is feasible and well tolerated in populations such as those found in Northern Louisiana. Investigators will assess the impact of psilocybin-facilitated treatment on methamphetamine abstinence, craving, negative affect, cognitive function and quality of life. Components of the psilocybin experience will also be measured (persisting effects, quality of life, challenging experiences, etc). Investigators will assess feasibility and tolerability as rates of retention and challenging experiences, among other factors.

DETAILED DESCRIPTION:
This is an open-label pilot study evaluating the feasibility and tolerability of a single 25 mg psilocybin dose in promoting abstinence from methamphetamine. Participants will attend 10 to 12 study visits over a period of up to six months.

Participants will be recruited from a population receiving treatment for methamphetamine dependence at a local residential treatment facility. Recruitment will involve informative presentations to current clients and counselor-facilitated referrals based on provided inclusion criteria. Prescreening will utilize information collected by the treatment center during the client's admission process.

Individuals who meet prescreening criteria will be invited to an in-person screening visit, conducted after obtaining informed consent. The screening visit will include a clinical review, a detailed psychiatric interview, self-report questionnaires, a comprehensive medical history, and safety laboratory testing, including blood draws.

Once eligibility is confirmed, participants will proceed with study enrollment and complete baseline assessments, which will measure substance use, quality of life, and executive function. Three preparatory sessions will follow over a two-week period to establish trust and rapport between participants and session monitors, educate participants on the study protocol, and prepare them for the psilocybin session. Two preparatory sessions may be conducted via telehealth to enhance feasibility, while the third will be conducted in person with both the primary and secondary monitors present. A medical examination will be performed within the week preceding psilocybin administration.

Within a week of the third preparatory session, participants will attend a psilocybin administration session. Participants will arrive at the study location by 9:30 AM and undergo safety screenings, including breathalyzer testing, before psilocybin administration at approximately 10:00 AM. Participants will have been instructed to consume a low-fat breakfast prior to arrival. During the session, cardiovascular measures (e.g., heart rate, blood pressure) will be monitored upon arrival, hourly throughout the session, and as clinically indicated.

The psilocybin session, lasting approximately 6-8 hours, will be monitored by both the primary and secondary session monitors, ensuring that at least one individual is present with the participant at all times. At the conclusion of the session, participants will complete questionnaires assessing their subjective experiences. Participants will then be released into the care of treatment center staff, who will provide emotional support. Participants will also receive contact information for the primary monitor to access support if needed.

Post-session integration will include two telehealth sessions: the first within one day of the psilocybin session and the second approximately 7 days later (±3 days). These sessions will provide opportunities to discuss insights or challenges arising from the psilocybin experience, with an emphasis on promoting adaptive cognitive and behavioral changes.

Follow-up assessments will occur via telehealth at 30 and 60 days post-psilocybin, with an in-person assessment conducted at 120 days. The final visit will include a urine drug screen.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-65 at time of signing informed consent
* Identification of methamphetamine as drug of choice
* Score of at least 3 on the Severity of Dependence Scale
* Have been at the designated local treatment facility for at least 7 days
* Use of methamphetamine in the month preceding admission to the treatment center
* Desire to cease methamphetamine use as indicated by a goal of complete methamphetamine abstinence on the Thoughts about Abstinence questionnaire
* All English speakers, as all neuropsychological tasks will be given in English
* No prior psychedelic use or it will have been at least 3 years since their last use of a psychedelic
* Ability to attend two telehealth and one in person preparatory session appointments to establish comfort, trust and rapport between subjects and the research team and discuss the subjects' goals and aspirations with regard to the psilocybin administration.
* Ability to attend two integration sessions via telehealth and 3 follow-up assessments in person and via telehealth.
* Diagnosis of Stimulant Use Disorder - Amphetamine type on the MINI (Mini International Neuropsychiatric Interview), with no other substance dependence diagnoses other than nicotine or cannabis
* In acute remission from methamphetamine for at least 7 days prior to experimental drug administration as assessed by self-report and confirmed by urine drug screen (UDS) as well as the lack of any acute signs of intoxication on psychoactive drugs other than nicotine

Exclusion Criteria:

* Meeting criteria for substance dependence diagnoses other than methamphetamine (except nicotine and cannabis) as assessed by the MINI
* History of Hallucinogen Use Disorder or Hallucinogen Persisting Perceptive Disorder
* Women who are pregnant, plan to become pregnant, or are breast feeding
* Women who do not agree to engage in abstinence or are not using dual contraceptive methods at the time of enrollment and for the study duration
* Current hypertension (exceeding 140 systolic and 90 diastolic at resting as described below) at screening or during vitals taken pre-dosing
* Heart rate of less than 60 bpm and greater than 100 bpm at screening or during vitals taken pre-dosing
* QTc of less than 350 msec or more than 460 msec
* History of cardiovascular disease (other than controlled hypertension) or cerebral vascular disease
* Unstable medical or psychiatric conditions or disorders as determined at the discretion of the attending psychiatrist
* Clear diagnosis of schizophrenia or type 1 bipolar disorder (clear from confusion with drug-induced acute states)
* Having current or recent (last 6 months) suicidal ideation, assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
* Subjects currently taking medications on the prohibited medications list or that are unwilling/unable to cease medication
* History of significant brain injury or seizure disorder
* Inability to understand the informed consent, study purpose and procedures, or other study materials involved in the research study
* Those with moderate to severe hepatic impairment, as assessed by laboratory parameters.
* Plans to move away from Shreveport-Bossier area in the next 6 months
* Subjects whose laboratory blood tests demonstrate clinically significant abnormalities. Clinically acceptable ranges listed below:

  * Complete Blood Count (CBC) Red Blood Cell Count (RBC): 4.5 - 6.0 million cells/µL

Hemoglobin (Hb or Hgb):

* For men: 13.8 - 17.2 g/dL
* For women: 12.1 - 15.1 g/dL

Hematocrit (Hct):

* For men: 38.3% - 48.6%
* For women: 35.5% - 44.9% White Blood Cell Count (WBC): 4,500 - 11,000 cells/µL Platelet Count: 150,000 - 450,000 cells/µL

  * Blood Chemistry with Liver Function Tests Alanine Transaminase (ALT): 7 - 56 units/L Aspartate Transaminase (AST): 8 - 48 units/L Bilirubin (Total): 0.2 - 1.2 mg/dL
  * Renal Function Tests Blood Urea Nitrogen (BUN): 7 - 20 mg/dL Creatinine: 0.6 - 1.3 mg/dL
  * If there are abnormalities, or if the results are outside the normal reference ranges, the subject may be included only if the investigator judges the abnormalities or deviations from normal to not be clinically significant, or indicative of an unstable medical condition.

Prohibited Medications If subjects have a history of taking the following medications, they should be discontinued at least 5 half-lives prior to administering psilocybin.

* Medications that antagonize the serotonin 2A receptor
* Medications with serotonergic activity (e.g., SSRIs, SNRIs, efavirenz, lithium)
* Medications that inhibit UGT1A9 or UGT1A10 enzymes
* Monoamine Oxidase Inhibitors (MAOIs)
* Medications that inhibit aldehyde or alcohol dehydrogenase

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Participant retention rate | Screening, Visit #1
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | Baseline Assessments, Visit #2
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | Preparatory Session #1, Visit #3 (on study day (-)14; 14 days prior to dosing)
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | Preparatory Session #2, Visit #4 (on study day (-) 7; 7 days prior to dosing)
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | Preparatory Session #3, Visit #5 (on study day (-)3; 3 days prior to dosing)
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | Day of drug administration, Visit #6 (on study day 0)
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | 1-Day post drug administration integration session, Visit #7
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | 7-Day post drug administration integration session, Visit #8
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | 30-days post drug administration follow-up (Follow-up #1), Visit #9
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | 60-days post drug administration follow-up (Follow-up #2), Visit #10
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Participant retention rate | 120-days post drug administration follow-up (Follow-up #3), Visit #11 (Final visit)
  Description: Retention in the study will be assessed by measuring the percentage of study visits completed per participant.
  Measure:
  * Retention rate (percent of scheduled study visits completed by each participant).
Preliminary efficacy of psilocybin on methamphetamine abstinence | Screening, Visit #1
  Description: Methamphetamine abstinence will be assessed using both objective and self-reported substance use measures.
  Measure:
  * Urine drug screen results (positive/negative for methamphetamine).
Preliminary efficacy of psilocybin on methamphetamine abstinence | Day of drug administration, Visit #6 (on study day 0)
  Description: Methamphetamine abstinence will be assessed using both objective and self-reported substance use measures.
  Measure:
  * Urine drug screen results (positive/negative for methamphetamine).
Preliminary efficacy of psilocybin on methamphetamine abstinence | 120 days post drug administration (Follow up #3), Visit #11(final visit)
  Description: Methamphetamine abstinence will be assessed using both objective and self-reported substance use measures.
  Measure:
  * Urine drug screen results (positive/negative for methamphetamine).
Preliminary efficacy of psilocybin on methamphetamine abstinence | Screening, Visit #1
  Description: Methamphetamine abstinence will be assessed using both objective and self-reported substance use measures.
  Measure:
  * Timeline Followback (TLFB): Self-reported days of methamphetamine use in the past 30 days.
Preliminary efficacy of psilocybin on methamphetamine abstinence | 30 day post drug administration (Follow up #1), Visit #9
  Description: Methamphetamine abstinence will be assessed using both objective and self-reported substance use measures.
  Measure:
  * Timeline Followback (TLFB): Self-reported days of methamphetamine use in the past 30 days.
Preliminary efficacy of psilocybin on methamphetamine abstinence | 60 day post drug administration (Follow up #2), visit #10
  Description: Methamphetamine abstinence will be assessed using both objective and self-reported substance use measures.
  Measure:
  * Timeline Followback (TLFB): Self-reported days of methamphetamine use in the past 30 days.
Preliminary efficacy of psilocybin on methamphetamine abstinence | 120 days post drug administration (Follow up #3), visit #11
  Description: Methamphetamine abstinence will be assessed using both objective and self-reported substance use measures.
  Measure:
  * Timeline Followback (TLFB): Self-reported days of methamphetamine use in the past 30 days.
Mystical experiences associated with psilocybin administration | Day of drug administration, Visit #6 (on study day 0)
  Description: The subjective effects of psilocybin will be assessed using validated self-report questionnaires.
  Measure:
  * Mystical Experience Questionnaire (MEQ-30): Total score range = 0-150; higher scores indicate a more intense mystical experience.
Challenging experiences associated with psilocybin administration | Day of drug administration, Visit #6 (on study day 0)
  Description: The subjective effects of psilocybin will be assessed using validated self-report questionnaires.
  Measure:
  * Challenging Experience Questionnaire (CEQ): Total score range = 0-200; higher scores indicate a more challenging experience.
Physiological responses to psilocybin administration | Baseline - Visit #2
  Description: The physiological effects of psilocybin will be monitored using cardiovascular measures collected before, during, and after drug administration.
  Measure:
  * Heart rate (beats per minute).
Physiological responses to psilocybin administration | Preparatory Session #3, Visit #5 (on study day (-)3; 3 days prior to dosing)
  Description: The physiological effects of psilocybin will be monitored using cardiovascular measures collected before, during, and after drug administration.
  Measure:
  * Heart rate (beats per minute).
Physiological responses to psilocybin administration | Day of drug administration(hourly) - Visit #6 (on study day 0)
  Description: The physiological effects of psilocybin will be monitored using cardiovascular measures collected before, during, and after drug administration.
  Measure:
  * Heart rate (beats per minute).
Physiological responses to psilocybin administration | Post-session monitoring day of drug administration - Visit #6 (on study day 0)
  Description: The physiological effects of psilocybin will be monitored using cardiovascular measures collected before, during, and after drug administration.
  Measure:
  * Heart rate (beats per minute).
Physiological responses to psilocybin administration | Baseline - Visit #2
  Description: The physiological effects of psilocybin will be monitored using cardiovascular measures collected before, during, and after drug administration.
  Measure:
  * Blood pressure (systolic/diastolic, mmHg).
Physiological responses to psilocybin administration | Preparatory Session #3, Visit #5 (on study day (-)3; 3 days prior to dosing)
  Description: The physiological effects of psilocybin will be monitored using cardiovascular measures collected before, during, and after drug administration.
  Measure:
  * Blood pressure (systolic/diastolic, mmHg).
Physiological responses to psilocybin administration | Day of drug administration(hourly) - Visit #6 (on study day 0)
  Description: The physiological effects of psilocybin will be monitored using cardiovascular measures collected before, during, and after drug administration.
  Measure:
  * Blood pressure (systolic/diastolic, mmHg).
Physiological responses to psilocybin administration | Post-session monitoring day of drug administration - Visit #6 (on study day 0)
  Description: The physiological effects of psilocybin will be monitored using cardiovascular measures collected before, during, and after drug administration.
  Measure:
  * Blood pressure (systolic/diastolic, mmHg).

SECONDARY OUTCOMES:
Effects of psilocybin on quality of life | Baseline assessment, visit #2
  Description: Quality of life will be assessed using a validated self-report questionnaire.
  Measure:
  * Quality of Life Questionnaire (QOL): Score range = 14-70; higher scores indicate greater life satisfaction.
Effects of psilocybin on quality of life | 30 day post drug administration (Follow up #1), Visit #9
  Description: Quality of life will be assessed using a validated self-report questionnaire.
  Measure:
  * Quality of Life Questionnaire (QOL): Score range = 14-70; higher scores indicate greater life satisfaction.
Effects of psilocybin on quality of life | 60 day post drug administration (Follow up #2), Visit #10
  Description: Quality of life will be assessed using a validated self-report questionnaire.
  Measure:
  * Quality of Life Questionnaire (QOL): Score range = 14-70; higher scores indicate greater life satisfaction.
Effects of psilocybin on quality of life | 120 days post drug administration (Follow up #3), Visit #11
  Description: Quality of life will be assessed using a validated self-report questionnaire.
  Measure:
  * Quality of Life Questionnaire (QOL): Score range = 14-70; higher scores indicate greater life satisfaction.
Effects of psilocybin on negative affect | Baseline assessment, Visit #2
  Description: Symptoms of depression, anxiety, and stress will be assessed using a validated self-report scale.
  Measure:
  * Depression Anxiety and Stress Scale (DASS-21): Score range = 0-126; higher scores indicate more severe negative affect.
Effects of psilocybin on negative affect | 30 day post drug administration (Follow up #1), Visit #9
  Description: Symptoms of depression, anxiety, and stress will be assessed using a validated self-report scale.
  Measure:
  * Depression Anxiety and Stress Scale (DASS-21): Score range = 0-126; higher scores indicate more severe negative affect.
Effects of psilocybin on negative affect | 60 day post drug administration (Follow up #2), visit #10
  Description: Symptoms of depression, anxiety, and stress will be assessed using a validated self-report scale.
  Measure:
  * Depression Anxiety and Stress Scale (DASS-21): Score range = 0-126; higher scores indicate more severe negative affect.
Effects of psilocybin on negative affect | 120 days post drug administration (Follow up #3), Visit #11
  Description: Symptoms of depression, anxiety, and stress will be assessed using a validated self-report scale.
  Measure:
  * Depression Anxiety and Stress Scale (DASS-21): Score range = 0-126; higher scores indicate more severe negative affect.

OTHER OUTCOMES:
Effects of psilocybin on cognitive flexibility | Baseline, visit #2
  Description: Cognitive flexibility will be assessed using a neuropsychological test that measures executive function and task-switching ability.
  Measure:
  * Trail Making Test (TMT Part B): Time to completion (seconds); shorter time indicates better executive function.
Effects of psilocybin on cognitive processing speed | 120 days post-drug administration (Follow Up #3), Visit #11.
  Description: Cognitive processing speed will be assessed using a standardized neuropsychological task.
  Measure:
  * Digit Symbol Substitution Task (DSST): Number of correct responses in 90 seconds; higher scores indicate better cognitive processing speed.
Effects of psilocybin on inhibitory control | Baseline, visit #2
  Description: Inhibitory control will be assessed using a validated cognitive task that measures response inhibition.
  Measure:
  * Stroop Color and Word Task: Reaction time (milliseconds); shorter reaction times indicate better inhibitory control.
Effects of psilocybin on inhibitory control | 120 days post-drug administration (Follow Up #3), Visit #11
  Description: Inhibitory control will be assessed using a validated cognitive task that measures response inhibition.
  Measure:
  * Stroop Color and Word Task: Reaction time (milliseconds); shorter reaction times indicate better inhibitory control.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin S Murnane, PhD, Principal Investigator — Louisiana State University Health Science Center Shreveport
Locations (1):
- LSU Health Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No